CLINICAL TRIAL: NCT04610398
Title: Perioperative Dexamethasone Reduces Postoperative Pain and Nausea After Hip Arthroscopy- a Double-blinded Placebo Controlled RCT
Brief Title: Perioperative Dexamethasone Reduces Postoperative Pain and Nausea After Hip Arthroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEXA and HAS
Record Dates: First submitted 2020-10-06; First posted 2020-10-30 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Pain, Postoperative; Nausea, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone group (Active Comparator): The patients in the dexamethasone group will receive 12mg dexamethasone (Fortecortin ®) intravenously 15-60 minutes prior to surgery while in general anasthesia as well as 12mg dexamethasone intravenously (Fortecortin®) on the first postoperative day at approx. 8.00a.m. by the investigators.
  Interventions: Drug: Dexamethasone 4mg
- Placebo/ Control group (Placebo Comparator): The patients will not receive any additional drugs preoperatively. A 0.9% NaCl Solution (NaCl B. Braun Inf Lös 0.9 % 250ml Ecoflac plus®) will be administered at approx. 8.00 a.m. on the first postoperative day by the investigators.
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Dexamethasone 4mg — s. arm/group description
  Other Names: Fortecortin Inject (Merck (Switzerland))
  Arms: Dexamethasone group
Drug: NaCl 0.9% — s. arm/group description
  Other Names: NaCL Braun (B.Braun Medical)
  Arms: Placebo/ Control group

SUMMARY:
The purpose of this study is to assess the effect of Dexamethasone on postoperative pain and nausea after hip arthroscopy.

DETAILED DESCRIPTION:
Hip arthroscopy (HAS) is a standard procedure with good mid and long-term results. Postoperative pain is a great concern and postoperative pain management of great importance. High demand for opiates and the associated side effects especially nausea limit the postoperative rehabilitation.

Promising results to reduce postoperative pain and nausea have been achieved by perioperative dexamethasone, which has a strong anti-inflammatory effect reducing pain and inflammation as well as a strong anti-emetic effect, especially in total hip replacement.

It is our goal to compare the effect of perioperative intravenous dexamethasone (3x 4mg Amp. Fortecortin =12mg prior to surgery and 3x4mg Amp. Fortecortin = 12mg at 8.00am of the first postoperative day in 250ml saline solution) to a control group (placebo) (1x 250ml saline solution postoperative day 1 at 8.00am) regarding pain level, opiate consumption, postoperative nausea and patient satisfaction.

A double-blinded prospective randomized control trial including 60 patients receiving elective unilateral HAS will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * general anasthesia
  * Elective isolated unilateral HAS for any reason
  * No Prior hip surgery
  * Written informed consent as documented by signature (Appendix Informed Consent Form)
  * Competent German language skills

Exclusion Criteria:

* • Chronic pain patient, chronic lower back pain

  * Steroid or immunosuppressive drugs used within 6 months of surgery
  * Renal failure, hepatic failure
  * Relevant allergies
  * Pregnancy/ Breast feeding
  * Contraindications for Fortecortin treatment according to Swissmedic
  * Previous enrollment into the current study
  * Participation in another study with investigational drug within the 30 days preceding and during the present study
  * Known or suspected non-compliance, drug or alcohol abuse
  * Illness according to "Warnings and Precautions of Dexamethasone and NaCl"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain level | 6 hours postoperatively
  The VAS Pain score assesses pain Levels on a scale from 0 (no pain) to 10 (wost possible pain).
Postoperative pain level | 24 hours postoperatively
  The VAS Pain score assesses pain Levels on a scale from 0 (no pain) to 10 (wost possible pain).
Amount of opiates (morphinequivalent) consumed | 48 hours postoperatively
  We will assess the amount of Opiates the Patient needed due to the performed Surgery during the hospital stay.
Amount of anti-emetics consumed (Ondansetron) | 48 houts postoperatively
  We will assess the amount of mg of anti- emetic drugs (Ondansetron) the Patient required during the Hospital stay.

SECONDARY OUTCOMES:
Patient satisfaction as assessed by the revised American pain society patient outcome questionnaire | 6 hours postoperatively
  Patient satisfaction will be assessed by the revised American pain Society Patient Outcome questionnaire (APS-POQ-R).
Patient satisfaction as assessed by the revised American pain society patient outcome questionnaire | 24 hours postoperatively
  Patient satisfaction will be assessed by the revised American pain Society Patient Outcome questionnaire (APS-POQ-R).
Patient satisfaction as assessed by the revised American pain society patient outcome questionnaire | 48 hours postoperatively
  Patient satisfaction will be assessed by the revised American pain Society Patient Outcome questionnaire (APS-POQ-R).
Number of vomiting events | 48 hours postoperatively
  We will Count the number of vomiting Events postoperatively as a direct marker for postoperative Nausea.
Physical therapy milestones | 48 hours postoperatively
  Our patients will be instructed and perform different postoperative Rehabilitation steps including (first steps in the hallway, Walking up and down stairs, bicycle Ergometer)
Length of hospitalization | after 1 week
  The length of hospitalization will be obtained from the Patient Chart.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Zingg, MD, Principal Investigator — PI
Locations (1):
- Uniklinik Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
If requested the individual participant data will be made available to other researchers.

REFERENCES:
- [Derived] Kaiser D, Hoch A, Dimitriou D, Groeber T, Bomberg H, Aguirre JA, Eichenberger U, Zingg PO. Perioperative Intravenous Dexamethasone Significantly Reduces Postoperative Opioid Requirement and Nausea After Unilateral Elective Hip Arthroscopy: A Randomized Double-blinded Placebo-controlled Trial. Am J Sports Med. 2024 Apr;52(5):1165-1172. doi: 10.1177/03635465241232157. Epub 2024 Mar 8. PMID 38456291